CLINICAL TRIAL: NCT02699606
Title: A Phase 2a Study to Evaluate The Clinical Efficacy of JNJ-42756493, A Pan-Fibroblast Growth Factor Receptor (FGFR) Tyrosine Kinase Inhibitor, In Asian Patients With Advanced Non-Small-Cell Lung Cancer, Urothelial Cancer, Gastric Cancer, Esophageal Cancer Or Cholangiocarcinoma
Brief Title: A Study to Evaluate the Clinical Efficacy of JNJ-42756493 (Erdafitinib), A Pan-Fibroblast Growth Factor Receptor (FGFR) Tyrosine Kinase Inhibitor, In Asian Participants With Advanced Non-Small-Cell Lung Cancer, Urothelial Cancer, Esophageal Cancer Or Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108120; 42756493LUC2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Neoplasm
Keywords: Tumor; Fibroblast Growth Factor Receptor (FGFR); Non-Small Cell Lung Cancer (NSCLC); Erdafitinib; Urothelial Cancer; Esophageal Cancer; Cholangiocarcinoma
MeSH Terms: conditions — Neoplasms; Acrocephalosyndactylia; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Cholangiocarcinoma | interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Erdafitinib (Experimental): Participants will receive a 8 milligram (mg) starting dose once daily with option to up-titrate to 9 mg on a 28-day cycle. The dose of study drug may be modified, delayed, or terminated based on guidelines provided in the protocol.
  Interventions: Drug: Erdafitinib

INTERVENTIONS:
Drug: Erdafitinib — Participants will receive 8 mg of erdafitinib, once daily with option to up-titrate to 9 mg.
  Other Names: JNJ-42756493

SUMMARY:
The primary purpose of this study is to evaluate objective response rate (ORR) as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of erdafitinib in a molecularly-defined subset of Asian participants with non-small-cell lung cancer (NSCLC), urothelial cancer, esophageal cancer and cholangiocarcinoma.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter, phase 2 study to evaluate the clinical efficacy, safety and pharmacokinetics of erdafitinib in Asian participants with advanced NSCLC, urothelial cancer, esophageal cancer and cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed, advanced or refractory tumors (there are no restriction on the total number of lines of prior therapies, but participant should have received at least 1 line of anti-cancer therapy [as per local standard of care]): Squamous and non-squamous non-small-cell lung cancer (NSCLC), esophageal cancer, urothelial cancer and cholangiocarcinoma
* Participants must meet the following molecular eligibility criteria (diagnosed at a central or local laboratory using either a tumor tissue based assay, which must indicate: at least one of following): a) fibroblast growth factor receptor (FGFR) gene translocations b) FGFR gene mutations c) Participants with evidence of FGFR pathway activation or other potential target/pathway inhibited by erdafitinib may also be considered and allowed for enrollment if supported by emerging biomarker data.
* The presence of measurable disease according to the RECIST, Version 1.1 Criteria, and documented disease progression as defined by RECIST (Version 1.1) at baseline
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1
* Female participants (of child bearing potential and sexually active) and male participants (with a partner of child bearing potential) must use medically acceptable methods of birth control. Male participants must use highly effective birth control measurements when sexually active and must not donate sperm
* Adequate bone marrow, liver, and renal function within the 14 days prior to Day 1 of Cycle 1 up until pre-dose of Cycle 1

Exclusion Criteria:

* Chemotherapy, targeted therapies, immunotherapy, or treatment with an investigational anticancer agent within 2 weeks or at least 5 half-lives of the drug whichever is longer up to a maximum of 4 weeks before the first administration of study drug. Localized palliative radiation therapy (but should not include radiation to target lesions) and ongoing luteinizing hormone-releasing hormone (LHRH) agonists, bisphosphonates and denosumab, are permitted
* Participants with persistent phosphate greater than (>) upper limit of normal (ULN) during Screening (within 14 days prior to Day 1 of Cycle 1 up until pre-dose of Cycle 1) and despite medical management of phosphate levels
* Participants taking medications known to have a significant risk of causing QTc prolongation and Torsades de Pointes. Participants who have discontinued any of these medications must have a wash-out period of at least 5 days or at least 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug
* Left ventricular ejection fraction (LVEF) less than (<) 50% as assessed by echocardiography (or multi-gated acquisition [MUGA]) performed at Screening
* Uncontrolled inter-current illness including, but not limited to, poorly controlled hypertension or diabetes, ongoing active infection requiring antibiotics, psychiatric illness, or at risk of gastrointestinal perforation as per investigators' assessment
* Received prior selective FGFR inhibitor treatment or RET inhibitor treatment, respectively according to the biomarker prescreening result, or if the participant has known allergies, hypersensitivity, or intolerance to Erdafitinib or its excipients
* Any corneal or retinal abnormality likely to increase risk of eye toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the date of the first dose of study drug until disease progression or death as assessed up to the last efficacy assessment for disease progression (approximately 2 years)
  Objective Response Rate (ORR) is defined as proportion of participants with best objective response of complete response (CR) or partial response (PR) based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) criteria.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From the date of the first dose of study drug until disease progression or death as assessed up to the last efficacy assessment for disease progression (approximately 2 years)
  Duration from the date of the first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death, whichever comes first.
Duration Of Response (DOR) | From the date of the first dose of study drug until disease progression or death as assessed up to the last efficacy assessment for disease progression (approximately 2 years)
  Duration of response is defined as the time from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death.
Disease Control Rate (DCR) | From the date of the first dose of study drug until disease progression or death as assessed up to the last efficacy assessment for disease progression (approximately 2 years)
  DCR defined as the proportion of participants with complete response [CR], partial response [PR], or greater than or equal to (>=) 6 weeks stable disease [SD]).
Overall Survival (OS) | From the date of the first dose of study drug until death, or withdrawal of consent or long-term extension (LTE) phase initiates, whichever occurs first (approximately 2 years)
  The OS is defined as the time from the date of first dose of study drug to date of death from any cause. If the participant is alive or the vital status is unknown, the participant will be censored at the date the participant will be last known to be alive.
Number of Participants With an Adverse Event | Screening up to end of study (approximately 2 years)
Plasma Concentration of Erdafitinib | Approximately up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- China (3):
  - Beijing
  - Harbin
  - Nanjing
- Seoul, South Korea
- Taiwan (2):
  - Kaohsiung City
  - Tainan

REFERENCES:
- [Derived] Park JO, Feng YH, Su WC, Oh DY, Keam B, Shen L, Kim SW, Liu X, Liao H, Qing M, Zhang C, Qian J, Tang X, Li P, Triantos S, Sweiti H. Erdafitinib in Asian patients with advanced solid tumors: an open-label, single-arm, phase IIa trial. BMC Cancer. 2024 Aug 13;24(1):1006. doi: 10.1186/s12885-024-12584-0. PMID 39138436